CLINICAL TRIAL: NCT01957020
Title: The Diagnostic Accuracy of Stereotactic Directional Vacuum-Assisted Breast Biopsy
Brief Title: Stereotactic Directional Vacuum-Assisted Breast Biopsy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200806017R
Record Dates: First submitted 2013-09-23; First posted 2013-10-08 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer; Stereotactic Directional Vacuum-assisted Breast Biopsy; Female; Adult Patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Stereotactic directional vacuum-assisted breast biopsy (ST DVAB) is a standard biopsy procedure for suspicious findings on mammograms in Western countries for more than 10 years [1-3], it has replaced the needle localization (NLOC) excisional biopsy for the lesions alike and was reported to feature a high sensitivity, very low delayed false-negative rate (less than 2%)[4,5]. Moreover, it causes less scarring, less psychologic stress to patients and less morbidity compared with needle localization excisional biopsy [6,7]. However, its sensitivity, accuracy has seldom been reported in Asian countries [8] , since most Asian women have different breast parenchyma pattern, different breast cancer prevalence. Therefore, we retrospectively reviewed outcomes of the two groups of patients receiving either ST DVAB or NLOC excisional biopsy, trying to investigate if ST DVAB can be an effective alternative to NLOC excisional biopsy in our country.

ELIGIBILITY:
Inclusion Criteria:

* The indication for ST DVAB was lesions with suspicious nature for malignancy seen on mammograms which biopsy is necessitated for tissue proof, or probably benign or benign appearing lesions seen on mammograms but patients or clinicians requested biopsy

Exclusion Criteria:

-

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: asymptomatic women with mammographic screening, and with suspicious findings on mammography.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The sensitivity of stereotactic vacuum assisted breast biopsy for breast cancer diagnosis | up to 5 years ( July 2008 to June 2013)
  the aforementioned outcome measure-"sensitivity"- is the probability of the stereotactic vaccum assisted breast biopsy can correctly diagnose the breast cancer. And according to statistical definition, it is defined as- for those breast cancer cases, how many of them can be correctly diagnosed by stereotactic breast biopsy.